CLINICAL TRIAL: NCT04908891
Title: A Comprehensive Assessment of Trunk, Scapula and Upper Limb in Neurological Patients. Reliability, Validity and Interrelatedness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Revalidatie & MS Centrum Overpelt (Other); Ziekenhuis Oost-Limburg (Other); National MS Center Melsbroek (Other); Jessa Hospital (Other)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Neuro-JR-001
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis; Stroke
MeSH Terms: conditions — Multiple Sclerosis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- persons with Multiple Sclerosis (Experimental)
  Interventions: Other: Clinical Scapular protocol (ClinScaP); Other: the prevalence of trunk, scapula and upper limb impairments.; Other: the interaction between trunk, scapula and upper limb impairments.
- Healthy controls (Active Comparator)
  Interventions: Other: Clinical Scapular protocol (ClinScaP)
- Stroke Patients (Active Comparator)
  Interventions: Other: the prevalence of trunk, scapula and upper limb impairments.; Other: the interaction between trunk, scapula and upper limb impairments.

INTERVENTIONS:
Other: Clinical Scapular protocol (ClinScaP) — the psychometric properties of two tests: Clinical Scapular protocol (ClinScaP) in PwMS and healthy controls.
  Arms: Healthy controls; persons with Multiple Sclerosis
Other: the prevalence of trunk, scapula and upper limb impairments. — To investigate the prevalence of trunk, scapula and upper limb impairments in PwMS and stroke patients.
  Arms: Stroke Patients; persons with Multiple Sclerosis
Other: the interaction between trunk, scapula and upper limb impairments. — To investigate the interaction between trunk, scapula and upper limb impairments in PwMS and stroke patients.
  Arms: Stroke Patients; persons with Multiple Sclerosis

SUMMARY:
The study aimed to provide insights in the coordination between trunk, shoulder and upper limb while reaching. Two main phases are present in this study:

In phase A: the psychometric properties of two tests: Clinical Scapular protocol (ClinScaP) in PwMS (Persons with Multiple Sclerosis) and healthy controls.

1. To investigate the test-retest reliability of the Clinical Scapular Protocol (ClinScaP) and the Reaching Performance Scale (RPS) in PwMS
2. To investigate the discriminative of the ClinScaP between PwMS and healthy controls
3. To investigate the discriminative of the RPS between PwMS and healthy controls
4. To investigate the concurrent validity of ClinScaP and RPS in PwMS, compared with upper limb dysfunction measurements.

   In phase B:
5. To investigate the prevalence of trunk, scapula and upper limb impairments in PwMS and stroke patients.
6. To investigate the interaction between trunk, scapula and upper limb impairments in PwMS and stroke patients.

ELIGIBILITY:
Inclusion criteria for all participants: Healthy controls, PwMS (Persons with Multiple Sclerosis) and stroke patients

* Age > 18 years
* Able to understand and execute the test instructions
* Able to sit on a chair with low back support for 10 minutes

Inclusion criteria specific for PwMS:

* Diagnosed with MS (Multiple Sclerosis) using McDonald criteria
* Able to move at least 1 out of 3 joints (wrist, elbow or shoulder): Medical Research Council score 3.

Inclusion criteria for stroke patients:

* First- ever single, unilateral (ischemic or hemorrhagic) stroke
* No apraxia or hemi spatial neglect
* Able to move at least 1 out of 3 joints of the affected upper limb (wrist, elbow or shoulder): Medical Research Council score 3.

Exclusion Criteria:

* Other medical conditions interfering with the upper limb function or trunk (orthopedic or rheumatoid impairment)
* Perceived pain in one of the upper limbs of more than 4/10 (Visual Analog Scale)
* Severe cognitive or visual deficits interfering with testing
* For the PwMS: a relapse or relapse-related treatment in the last month prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
The Reaching performance scale (RPS) | baseline
  The Reaching performance scale (RPS) evaluates 6 components during reaching to a cup. The first four components:
  1. trunk displacement,
  2. movement smoothness,
  3. shoulder movements, and
  4. elbow movements. The components are evaluated during reaching movements to targets placed close or far from the person. The 2 additional components globally rate
  5. the quality of prehension and
  6. the accomplishment of the task.
The Reaching performance scale (RPS) | Day 1
  The Reaching performance scale (RPS) evaluates 6 components during reaching to a cup. The first four components:
  1. trunk displacement,
  2. movement smoothness,
  3. shoulder movements, and
  4. elbow movements. The components are evaluated during reaching movements to targets placed close or far from the person. The 2 additional components globally rate
  5. the quality of prehension and
  6. the accomplishment of the task.
The clinical scapular protocol | Baseline
  The clinical scapular protocol consists of five items. A score is given between 0 and 2, based on observation of tilting and winging, shoulder girdle position (measuring acromial and pectoralis minor index and scapular distance test), scapular lateral rotation, maximal active humeral elevation, medial rotation test
The clinical scapular protocol | day 1
  The clinical scapular protocol consists of five items. A score is given between 0 and 2, based on observation of tilting and winging, shoulder girdle position (measuring acromial and pectoralis minor index and scapular distance test), scapular lateral rotation, maximal active humeral elevation, medial rotation test

SECONDARY OUTCOMES:
Trunk Impairment Scale | Baseline
  Trunk Impairment Scale used to measure static and dynamic sitting balance and trunk coordination in a sitting position.
Trunk Impairment Scale | day 1
  Trunk Impairment Scale used to measure static and dynamic sitting balance and trunk coordination in a sitting position.
Box and Block test | Baseline
  This test assess gross manual dexterity by grasping each time one block and transporting the block to the other side over a wooden panel for one minute, while sitting.
Box and Block test | day 1
  This test assess gross manual dexterity by grasping each time one block and transporting the block to the other side over a wooden panel for one minute, while sitting.
The Brunnström Fugl Meyer (BFM) | Baseline
  The Brunnström Fugl Meyer (BFM) used to measure motor control at the body functions and structures level. The upper limb section is applied: shoulder, elbow, forearm, wrist movements and grip.
The Brunnström Fugl Meyer (BFM) | day 1
  The Brunnström Fugl Meyer (BFM) used to measure motor control at the body functions and structures level. The upper limb section is applied: shoulder, elbow, forearm, wrist movements and grip.
The Action Research Arm Test (ARAT) | Baseline
  Action Research arm test, which assessed the patient's ability to handle objects varying in size, weight and shape. The Action Research Arm Test (ARAT) assess the ability to manipulate objects in different size, weight and shape and finally results in a maximum score of 57
The Action Research Arm Test (ARAT) | day 1
  Action Research arm test, which assessed the patient's ability to handle objects varying in size, weight and shape. The Action Research Arm Test (ARAT) assess the ability to manipulate objects in different size, weight and shape and finally results in a maximum score of 57
The Nine Hole Peg Test (NHPT) | baseline
  The Nine Hole Peg Test (NHPT) was used to assess manual dexterity by the time needed to place and remove nine pegs in a board.
The Nine Hole Peg Test (NHPT) | day 1
  The Nine Hole Peg Test (NHPT) was used to assess manual dexterity by the time needed to place and remove nine pegs in a board.
The Manual Ability Measure-36 (MAM-36) | baseline
  The Manual Ability Measure-36 (MAM-36) was used to assess perceived upper limb performance. The sum score is converted and resulted in a score between 0-100, with 100 as a perfect manual ability.
The Manual Ability Measure-36 (MAM-36) | day 1
  The Manual Ability Measure-36 (MAM-36) was used to assess perceived upper limb performance. The sum score is converted and resulted in a score between 0-100, with 100 as a perfect manual ability.
Arm Function in Multiple Sclerosis Questionnaire | Baseline
  : A Questionnaire Fatigue to evaluate the perceived performance of Arm Function in Multiple Sclerosis
Arm Function in Multiple Sclerosis Questionnaire | Day 1
  : A Questionnaire Fatigue to evaluate the perceived performance of Arm Function in Multiple Sclerosis
Active and passive range of motion of shoulder, elbow and wrist movement | Baseline
  Active and passive range of motion of shoulder, elbow and wrist movement is measured with a goniometer Safety Issue?: Yes/No
Active and passive range of motion of shoulder, elbow and wrist movement | Day 1
  Active and passive range of motion of shoulder, elbow and wrist movement is measured with a goniometer Safety Issue?: Yes/No
Modified Ashworth Scale | Baseline
  Spasticity is evaluated with Modified Ashworth Scale
Modified Ashworth Scale | day 1
  Spasticity is evaluated with Modified Ashworth Scale
Maximal hand grip strength test (HGS) | Baseline
  HGS was assessed with the Jamar digital HGD (the hand grip dynamometer). Each participant performed three maximum contractions of each hand on three handle positions progressing from first to third position.
Maximal hand grip strength HGS) | Day 1
  HGS was assessed with the Jamar digital HGD (the hand grip dynamometer). Each participant performed three maximum contractions of each hand on three handle positions progressing from first to third position.
Symbol digit modalities test | Baseline
  Information of processing speed with the Symbol digit modalities test
Symbol digit modalities test | Day 1
  Information of processing speed with the Symbol digit modalities test
Modified fatigue impact scale | Baseline
  : Fatigue is evaluated a questionnaire: the modified fatigue impact scale
Modified fatigue impact scale | Day 1
  : Fatigue is evaluated a questionnaire: the modified fatigue impact scale
National Institutes of Health Stroke Scale (NIHSS) | Baseline
  The National Institutes of Health Stroke Scale is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.[1] The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0
National Institutes of Health Stroke Scale (NIHSS) | Day 1
  The National Institutes of Health Stroke Scale is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.[1] The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0
10 Meter loop test (10MWT) | baseline
  The 10MWT assesses walking speed in meters per second over a short duration. (specific for stroke)
10 Meter loop test (10MWT) | Day 1
  The 10MWT assesses walking speed in meters per second over a short duration. (specific for stroke)
Modified Rankin Scale (MRS) | Baseline
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke
Modified Rankin Scale (MRS) | day 1
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Lamers, dr., Study Chair — Hasselt University
Locations (4):
- Belgium (4):
  - Ziekenhuis Oost-Limburg, Genk
  - Jessa Ziekenhuis- Campus St. Ursula, Herk-de-Stad
  - National MS Center Melsbroek, Melsbroek
  - Noorderhart MS & Revalidatie, Overpelt